CLINICAL TRIAL: NCT07219082
Title: Behavioral Safety and Fentanyl Education: BSAFE
Acronym: BSAFE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Francisco Department of Public Health (Other Government)
Responsible Party: Principal Investigator, Phillip Coffin, MD, MIA, Director, Substance Use Research, San Francisco Department of Public Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01DA064340-01 (NIH)
Record Dates: First submitted 2025-10-17; First posted 2025-10-21 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Drug Overdose; Drug Overdose Accidental
MeSH Terms: conditions — Drug Overdose

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BSAFE Counseling Intervention (Experimental): The BSAFE intervention will consist of three elements: motivational interviewing-based Counseling focused on a personalized plan to reduce risk for UFU and resultant overdose, (2) weekly text message Safety Reminders, and (3) Linkage to Care for managing stimulant use. The brief counseling intervention will utilize Motivational Interviewing and skills-building techniques to modify personal overdose risk behaviors.
  Interventions: Behavioral: BSAFE Intervention
- Attention Control (Placebo Comparator): Participants will watch 45 minute videos unrelated to the intervention as an attention control.
  Interventions: Behavioral: Attention control

INTERVENTIONS:
Behavioral: BSAFE Intervention — The intervention will include counseling sessions, reminder safety text messages, and linkage to care.
  Arms: BSAFE Counseling Intervention
Behavioral: Attention control — Attention control (videos)
  Arms: Attention Control

SUMMARY:
BSAFE is a randomized trial of a repeated-dose brief intervention to reduce overdose and risk behaviors among people who use stimulants who may have unintentional fentanyl use (UFU). It includes an established overdose education curriculum within an Informational-Motivation-Behavior (IMB) model. This study will test the efficacy of BSAFE vs attention-control.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older,
2. Reports intentional cocaine or methamphetamine use >15 of past 30 days,
3. Urine positive for cocaine or methamphetamine and negative for opioids/fentanyl prior to enrollment
4. Be able to provide the names of at least 2 persons who can consistently locate their whereabouts.

Exclusion Criteria:

1. Reports past 30-day intentional use of any opioid or ongoing use of an opioid antagonist (e.g., naltrexone)
2. Intends to leave area in coming year,
3. Unable to communicate in English or Spanish,
4. Any other condition that, in the PI's judgment, interferes with safe study participation or adherence to study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2030-01-15 (Estimated); Study Completion 2030-01-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of opioid overdose due to unintentional fentanyl use | 16 months
  Incidence of overdose will be measured by a composite measure of non-fatal and fatal overdose count collected by blinded assessors from Timeline Follow-Back (TLFB) every 4 months and vital record linkage for overdose fatalities.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip O Coffin, MD, MIA, Principal Investigator — San Francisco Department of Public Health
Locations (1):
- San Francisco Department of Public Health, San Francisco, California, United States